CLINICAL TRIAL: NCT04858295
Title: A Pilot Trial of the Feasibility of a Patient-Centered Mobile Health Self-Management Support Tool for Healthy Behaviors (SMART-HABITS) in Chronic Kidney Disease
Brief Title: Supporting Self-Management of Healthy Behaviors in Chronic Kidney Disease
Acronym: SMART-HABITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 832097; K23DK118198-03 (NIH)
Record Dates: First submitted 2021-03-31; First posted 2021-04-26 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Renal Insufficiency, Chronic; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Texting Arm (Active Comparator): Participants will receive automated text message reminders to check their blood pressure (BP) at least three days per week (participants will choose which days and times to receive reminders). Participants will transmit BP readings with text message to the Way to Health server. If a BP reading is not received within 3 hours, another reminder will be sent. Automated text message feedback will be sent with a tailored message. Participants will asked to set a daily step goal of at least 3,000 steps per day and transmit their step count information from their FitBit. Participants will be reminded once a day to sync their FitBit. Motivating messages will be sent weekly. After 4 weeks, and 8 weeks of the study, a usability survey will be sent. Weekly and daily feedback will be sent. At the conclusion of week 6, individuals will "crossover" and will continue for an additional 6 weeks using the opposite technology to communicate BP readings.
  Interventions: Device: Texting
- mHealth app Arm (Active Comparator): Participants randomized to the mHealth app (Omron Connect) arm will receive reminder messages to check their BP via push notifications from the Omron Connect app at least three times weekly. Upon receipt of the BP reading to the research platform from Omron Connect, participants will receive automatic tailored text message feedback similar to the texting arm. Participants will asked to set a daily step goal of at least 3,000 steps per day and transmit their step count information from their FitBit. Participants will be reminded once a day to sync their FitBit. Motivating messages will be sent weekly. After 4 weeks, and 8 weeks of the study, a usability survey will be sent. Weekly and daily feedback will be sent. At the conclusion of week 6, individuals will "crossover" and will continue for an additional 6 weeks using the opposite technology to communicate BP readings.
  Interventions: Device: mHealth app

INTERVENTIONS:
Device: Texting — The Way to Health platform is an automated information technology platform that integrates wireless devices, clinical trial randomization and enrollment processes, messaging (text, e-mail, voice), self-administered surveys, and secure data capture for research purposes. Way to Health has been used successfully in prior behavior intervention studies.
  Other Names: Way to Health; SMS Text
  Arms: Texting Arm
Device: mHealth app — Omron Connect app available on a participant's smartphone connects to the participant's home Omron blood pressure monitor via bluetooth technology. The Omron Connect app, which stores the blood pressure readings and provides reminders to the participant via push notifications also communicates with the Way to Health research platform via Internet connection.
  Other Names: Omron Connect; Smartphone application
  Arms: mHealth app Arm

SUMMARY:
The pilot cross-over study aims to examine the feasibility of a smartphone-based self-management supportive intervention, Supporting Self-Management of Healthy Behaviors (SMART-HABITS) in patients with chronic kidney disease (CKD) and hypertension. SMART-HABITS is a web-based application accessible on any device that has Internet access and utilizes a mobile health research platform (Way to Health) that links to wearable sensor smartphone applications such as FitBit and Omron Connect, to provide reminders, tailored feedback, and provide access to educational resources, and to community resources. The cross-over design is used to test preferences of using text message or a smartphone app to communicate blood pressure readings.

DETAILED DESCRIPTION:
The pilot study aims to examine the feasibility, as measured by adoption, adherence, and acceptance, of a smartphone-based self-management supportive intervention, Supporting Self-Management of Healthy Behaviors (SMART-HABITS) in patients with chronic kidney disease (CKD) and hypertension. SMART-HABITS is a web-based application accessible on any device that has Internet access and utilizes the mobile health research platform to provide the components of the intervention: a) text message reminders (Arm 1), b) text message tailored feedback (Arm 1 and 2), c) positive affirmation text messages (Arms 1 and 2), d) access to educational resources, community resources, CKD patient forums (Arms 1 and 2), e) option to select a accountability partner to share reminders and feedback (Arms 1 and 2). SMART-HABITS encompasses multiple behavior change techniques and is centered on the Health Belief Model and the Social Cognitive Theory. SMART-HABITS will deliver reminder text messages to a participant's smartphone to perform blood pressure self-monitoring in one arm and encourage an increase in walking activity both arms. The Omron Connect app will deliver the reminder notifications to check blood pressure and will deliver the BP readings to research platform (in the non-texting arm). After blood pressure measurements and daily step counts are remotely transmitted from the smartphone to mobile health research platform server, tailored feedback will be provided via text message). Additionally, intermittent positive affirmation messages will also be sent to participants to encourage engagement in the behaviors. Within the SMART-HABITS web-based application, there will be a participant portal that will provide access to links to community resources, educational links about CKD, and a display of adherence to behaviors and data transmission. At the beginning and end of the study, questionnaires will be completed to assess patient-reported outcomes, which will serve as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with hypertension (treated with three or less anti-hypertensive medications) and chronic kidney disease stage 3 or 4 managed in participating nephrology practices
* have a smartphone that they are willing to carry with them the majority of the time while enrolled in the study
* able to comprehend English,
* have ability to walk.
* mean blood pressure of <=180/100 mmHg from historical blood pressure readings in the electronic medical record
* able and willing to provide informed consent

Exclusion Criteria:

* inability to provide consent or read or speak English
* had MI or stroke within the previous six months,
* diagnosis of dementia or cognitive impairment
* inability to walk
* already participating in another physical activity study
* belong to vulnerable population
* likely to receive a kidney transplant within 1 month of enrollment into the trial
* living in a long-term care or rehabilitation institution
* likely to have their care transferred to another facility outside participating clinic areas during the course of the study
* planning to travel or live consecutively out of the country for more than one month
* participating in another intervention trial,
* hypertension not managed by the nephrologist in the clinic
* prescribed more than three anti-hypertensive medications (i.e. resistant hypertension),
* any other reason they do not expect to be able to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schrauben, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Derived] Schrauben SJ, Park D, Amaral S, Purcell A, Zhang S, Kearney M, Bilger A, Feldman HI, Dember LM. Supporting Self-Management of Healthy Behaviors in Chronic Kidney Disease and Hypertension: The Supporting Self-Management of Healthy Behaviors Pilot Randomized Trial. Clin J Am Soc Nephrol. 2024 Sep 1;19(9):1109-1118. doi: 10.2215/CJN.0000000000000492. Epub 2024 Jul 2. PMID 38954482

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 of 221 screened participants were randomized. Of those not randomized 40 declined to participate, and 134 did not meet inclusion criteria.
Groups:
- Text Message and Then mHealth App Arm: Participants will receive automated text message reminders to check their blood pressure (BP) at least three days per week (participants will choose which days and times to receive reminders). Participants will transmit BP readings with text message to the Way to Health server. If a BP reading is not received within 3 hours, another reminder will be sent. Automated text message feedback will be sent with a tailored message. Participants will asked to set a daily step goal of at least 3,000 steps per day and transmit their step count information from their FitBit. Participants will be reminded once a day to sync their FitBit. Motivating messages will be sent weekly. After 4 weeks, and 8 weeks of the study, a usability survey will be sent. Weekly and daily feedback will be sent. At the conclusion of week 6, individuals will "crossover" and will continue for an additional 6 weeks using the mHealth app to communicate BP readings.
  Texting: The Way to Health platform is an automated information technology platform that integrates wireless devices, clinical trial randomization and enrollment processes, messaging (text, e-mail, voice), self-administered surveys, and secure data capture for research purposes. Way to Health has been used successfully in prior behavior intervention studies.
- mHealth App Then Texting Arm: Participants randomized to the mHealth app (Omron Connect) arm will receive reminder messages to check their BP via push notifications from the Omron Connect app at least three times weekly. Upon receipt of the BP reading to the research platform from Omron Connect, participants will receive automatic tailored text message feedback similar to the texting arm. Participants will asked to set a daily step goal of at least 3,000 steps per day and transmit their step count information from their FitBit. Participants will be reminded once a day to sync their FitBit. Motivating messages will be sent weekly. After 4 weeks, and 8 weeks of the study, a usability survey will be sent. Weekly and daily feedback will be sent. At the conclusion of week 6, individuals will "crossover" and will continue for an additional 6 weeks using the text message to communicate BP readings.
  mHealth app: Omron Connect app available on a participant's smartphone connects to the participant's home Omron blood pressure monitor via bluetooth technology. The Omron Connect app, which stores the blood pressure readings and provides reminders to the participant via push notifications also communicates with the Way to Health research platform via Internet connection.
Period: All Study Participants
Arm/Group | Text Message and Then mHealth App Arm | mHealth App Then Texting Arm
Started | 23 | 24
Received Intervention | 23 | 23
Completed | 22 | 21
Not Completed | 1 | 3
Period: First Intervention (6 Weeks)
Arm/Group | Text Message and Then mHealth App Arm | mHealth App Then Texting Arm
Started | 23 | 24
Received Intervention | 23 | 23
Completed | 23 | 21
Not Completed | 0 | 3
Period: Second Intervention (6 Weeks)
Arm/Group | Text Message and Then mHealth App Arm | mHealth App Then Texting Arm
Started | 23 | 21
Completed | 22 | 21
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomized in the cross-over trial.
Groups:
- All Study Participants: All study participants were randomized to two approaches to communicate home blood pressure readings, with an mHealth app (Omron Connect) for 6 weeks and with text messages for the alternate 6 weeks.
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [52 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian/Alaskan Native | 1
  Race/Ethnicity: Asian | 2
  Race/Ethnicity: Black or African American | 21
  Race/Ethnicity: White or Caucasian | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47
Highest Level of Education [Count of Participants; unit: Participants]
  ≤High school | 6
  Some college | 14
  College or more | 27
Employment Status [Count of Participants; unit: Participants]
  Employed | 16
  Not Employed | 4
  Retired | 20
  Unable to work/disabled | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Adoption
Description: Composite outcome determined by participant retention rate, any use of the SMART-HABITS dashboard; Good adoption will be determined by greater than or equal to 70 percent of those retained in the study, and greater than or equal to 70 percent of those enrolled who actually used SMART-HABITS dashboard/web app as measured by data usage statistics.
Time Frame: Collected throughout study (12 weeks)
Population: Participants randomized to intervention sequence.
Measure: Count of Participants; unit: Participants
Groups:
- Per Intervention: Text Message: Participants assigned to self-report home blood pressure readings for 6 weeks with text message.
- Per Intervention: mHealth App: Participants assigned to report home blood pressure readings for 6 weeks with a smartphone app paired with a Bluetooth-capable blood pressure machine.
Arm/Group | Per Intervention: Text Message | Per Intervention: mHealth App
Number analyzed (Participants) | 47 | 47
Participants
  Retention | 44 | 42
  Any use of SMART-HABITS | 18 | 22

2. Primary Outcome: Feasibility: Adherence
Description: Determined by the number of blood pressure assessments and step counts performed divided by the number of assessments recommended. Good adherence will be determined by greater than or equal to 70 percent performed out of the recommended.
Time Frame: Collected throughout study (12 weeks)
Population: Participants receiving intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Texting Arm | mHealth App Arm
Number analyzed (Participants) | 47 | 47
Participants
  Adherence to 3 or more BP transmissions per week | 36 | 30
  Adherence to 5 or more daily step count transmissions per week | 43 | 43

3. Primary Outcome: Feasibility: Change in Acceptability of mHealth From Baseline (Pre-study) and 12 Weeks (Post-study)
Description: Determined through change in pre- and post-study scores on the three attitude statements toward mHealth, entitled Attitudes Toward Mobile Phone-Based Health Monitoring. Answers reported on 5-point Likert scale ranging from 1= strongly disagree, 2=disagree, 3=neither disagree or agree, 4=agree, to 5 = strongly agree (total range 3-15), with higher scores indicating better acceptability.
  If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) so all participants had completed both arms after the crossover, so all study participants who completed the end of study questionnaire were analyzed together regardless of arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
score on a scale | 12 [10 to 14]

4. Primary Outcome: Feasibility: Acceptability of SMART-HABITS
Description: Determined through satisfactory ratings on the System Usability Scale Survey (range is 0-100 with score above 68 considered adequate usability).
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: participants completing questionnaire at 4-weeks, 8 weeks and 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Text Message First (at 4 Weeks): Study participants randomized to text message at 4 weeks
- mHealth App (at 4 Weeks): Study participants randomized to mHealth app first who completed survey.
- Text Message Then mHealth App (at 8 Weeks): Study participants randomized to text message first and crossed over at 6 weeks to mHealth app who completed survey at 8 weeks.
- mHealth App Then to Text Message (at 8 Weeks): Study participants randomized to mHealth app first and crossed over at 6 weeks to text message who completed usability survey at 8 weeks.
- 12 Week Usability Survey of Those Who Received Text Message Arm First: Study participants randomized to text message first and crossed over at 6 weeks to mHealth app who completed survey at 12 weeks.
- 12 Week Usability Survey of Those Two Received mHealth Arm First: Study participants randomized to mHealth app first and crossed over at 6 weeks to text message who completed usability survey at 12 weeks.
Arm/Group | Text Message First (at 4 Weeks) | mHealth App (at 4 Weeks) | Text Message Then mHealth App (at 8 Weeks) | mHealth App Then to Text Message (at 8 Weeks) | 12 Week Usability Survey of Those Who Received Text Message Arm First | 12 Week Usability Survey of Those Two Received mHealth Arm First
Number analyzed (Participants) | 23 | 24 | 23 | 16 | 23 | 24
score on a scale | 77 (16.2) | 64.5 (19.7) | 70.1 (14.8) | 65.9 (19.4) | 71.6 (16.4) | 65.6 (21.7)

5. Secondary Outcome: Change in CKD Knowledge Scores From Baseline (Pre-study) and 12 Weeks (Post-study)
Description: Determined by change in pre-pilot and post-pilot scores on responses regarding CKD knowledge using the 28-question Kidney Knowledge Survey (KiKS). The survey score is defined the percentage correct responses to each answered question divided by the total, total range 0-100%. Higher percentages indicate better knowledge.
  If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) so all participants had completed both arms of the crossover, so all study participants who completed the end of study questionnaire were analyzed together regardless of arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 38
score on a scale | 66.7 [66.6 to 66.8]

6. Secondary Outcome: Change in Self-Efficacy of Managing Chronic Disease Scores From Baseline (Pre-study) and 12 Weeks (Post-study)
Description: Determined by change in pre-pilot and post-pilot scores on responses regarding self-efficacy using the Self-Efficacy for Managing Chronic Disease 6-Item Scale. Answer range from 1 = not at all confident to 10= totally confident, with higher scores indicating higher self-efficacy.
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) so all participants had completed both arms of the crossover, so all study participants who completed the end of study Self-Efficacy for Management Chronic Disease survey were analyzed together regardless of arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 38
score on a scale | 7.8 [6.95 to 8.65]

7. Secondary Outcome: Change in Self-Management Scores From Baseline (Pre-study) and 12 Weeks (Post-study)
Description: Determined by change in pre-pilot and post-pilot scores on responses regarding self-management using the Partners in Health Scale for Chronic Condition Self-Management (11 items). Answers range on a linear scale provided: very good=0, 1, 2, 3, 4=satisfactory, 5, 6, 7, 8= very poor. Total range of scores 0-88, with higher scores indicating better self-management.
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) so all participants had completed both arms of the crossover, so all study participants who completed the end of study Partners in Health Scale for Chronic Condition Self-management were analyzed together regardless of arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
score on a scale | 72 [64.5 to 79.5]

8. Secondary Outcome: Change in eHealth Literacy Scores From Baseline (Pre-study) and 12 Weeks (Post-study)
Description: Determined by change in pre-pilot and post-pilot scores on responses regarding eHealth literacy Scale (eHEALS). eHEALS consists of eight questions with 5 response options on a Likert-scale, and scored as a cumulative score of the eight questions (total range 8-40) with higher scores indicating better eHealth literacy (a score of ≥32 is considered to be adequate eHealth literacy).
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) so all participants had completed both arms of the crossover, so all study participants who completed the end of study eHealth Literacy Scale (eHEALS) were analyzed together regardless of arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
score on a scale | 30.5 [27.6 to 33.4]

9. Secondary Outcome: Change in Kidney Disease Quality of Life From Baseline (Pre-study) and 12 Weeks (Post-study)
Description: Determined by change in pre-pilot and post-pilot scores on responses regarding disease-related quality of life using the Kidney Disease Quality of Life 36-item survey (KDQOL-36). Scores are reported separately for each of the three KDQOL-36 subscales: Symptoms and Problems (12 items), Burden of Kidney Disease (4 items), and Effects of Kidney Disease (8 items); all items have 5 response options. Each sub-scale scores are transformed to 0 to 100 with higher scores indicating better quality of life.
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) so all participants had completed both arms of the crossover, so all study participants who completed the end of study KDQOL-36 were analyzed together regardless of arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
score on a scale
  Burden of Kidney Disease | 77.5 (23.9)
  Effects of Kidney Disease | 83.4 (24.4)
  Symptoms/Problems | 85.9 (21.4)

10. Secondary Outcome: Effectiveness of Home Monitoring of BP
Description: Mean systolic blood pressure after 4, 8, and 12 weeks
Time Frame: 4, 8, and 12 weeks
Population: All study participants randomized.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Per Intervention: Text Message: Participants self-report home blood pressure measures with text message for 6 weeks.
- Per Intervention: mHealth App: Participants automatically report home blood pressure measures with smartphone app connected to Bluetooth-enabled blood pressure machine for 6 weeks.
Arm/Group | Per Intervention: Text Message | Per Intervention: mHealth App
Number analyzed (Participants) | 47 | 47
mmHg
  SBP at 4 weeks | 125 (9) | 130 (12)
  SBP at 8 weeks | 125 (10) | 129 (12)
  SBP at 12 weeks | 126 (9) | 129 (14)

11. Secondary Outcome: Effectiveness of Step Monitoring
Description: Mean step count in first week, and after 4, 8, and 12 weeks.
Time Frame: 4, 8, and 12 weeks
Population: The outcome measure was collected on daily basis regardless of BP communication arm at 4-, 8-, and 12 weeks.
Measure: Mean (Standard Deviation); unit: daily steps
Groups:
- Per Intervention: Mhealth App: Participants assigned to report home blood pressure readings for 6 weeks with mhealth App.
Arm/Group | Per Intervention: Text Message | Per Intervention: Mhealth App
Number analyzed (Participants) | 47 | 47
daily steps
  Daily steps in week 1 | 6846 (3902) | 5897 (3541)
  Daily steps in week 4 | 6758 (4142) | 6250 (3400)
  Daily steps in week 8 | 7387 (4614) | 6106 (4081)
  Daily steps in week 12 | 6515 (3994) | 6153 (3282)

12. Secondary Outcome: Maintenance
Description: Determined by transmitting at least one BP monitored reading or daily step count each week.
Time Frame: 12 weeks
Population: The outcome measure was collected at 12 weeks (end of study) regardless of arm and BP communication mode so participants were analyzed regardless of arm.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Participants | 43

13. Secondary Outcome: Implementation Issues
Description: Qualitative reports describing adaptions that were made to the SMART-HABITS program in response to participant feedback, including descriptions of alterations that were made to the schedule of reminders and messaging content. Participant feedback data will be collected with field notes from verbal conversations and textual data from email and text messages.
Time Frame: 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Reach: Qualitatively Similar Frequency of the Sex Distribution of Participants in the Study at the Time of Randomization vs. Published Information on the US General Population With Chronic Kidney Disease Stage 3 and 4 With Hypertension
Description: Sex frequency of randomized participants compared to the published sex frequency of the US population with CKD (female approximately 55%)
Time Frame: At the time of randomization
Population: Compare the frequency of demographic characteristic of all participants randomized to that of published frequency of demographics of the US population with CKD
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Participants
  Female | 23
  Male | 24

15. Secondary Outcome: Reach: Qualitatively Similar Frequency (Percentage) of the Race Group Distribution of Randomized Participants vs. US General Population With Chronic Kidney Disease Stage 3 and 4 With Hypertension
Description: Frequency of race groups (Black, White other) of participants at time of randomization compared to the approximate frequency---- of the US population with CKD (black race group = 18%, white race group = 75%)
Time Frame: At time of randomization
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Participants
  Black | 21
  White | 23
  American Indian/Alaskan Native | 1
  Asian | 2

16. Secondary Outcome: Reach: Qualitatively Similar Frequency (Percentage) of the Ethnic Group Distribution of Randomized Participants vs. US General Population With Chronic Kidney Disease Stage 3 and 4 With Hypertension
Description: Determined by the comparison of ethnicity (Hispanic, Non-Hispanic) frequency (percentage) of the randomized participants compared to ethnicity frequency of the general population with chronic kidney disease stage in the United States (Hispanic = ~13%).
Time Frame: Enrolled and randomized
Population: Participants who were randomized
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Participants
  Hispanic ethnicity | 1
  Non-Hispanic | 46

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire study duration (12 weeks) for each participant.
Arm/Group | Texting Arm | mHealth App Arm
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT04858295/Prot_SAP_ICF_000.pdf